CLINICAL TRIAL: NCT06594159
Title: A Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of LY4065967, to Evaluate the Effect of LY4065967 on the Pharmacokinetics of Rosuvastatin in Healthy Japanese Participants
Brief Title: A Study of LY4065967 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18815; J4X-JE-LWCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A and B-Double-blinded Part A3 and D-Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY4065967 Part A (Experimental): A single dose of LY4065967 administered orally
  Interventions: Drug: LY4065967
- Placebo Part A (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- LY4065967 Part B (Experimental): Multiple doses of LY4065967 administered orally
  Interventions: Drug: LY4065967
- Placebo Part B (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- LY4065967 and Rosuvastatin Part D (Experimental): LY4065967 and Rosuvastatin administered orally
  Interventions: Drug: LY4065967; Drug: Rosuvastatin

INTERVENTIONS:
Drug: LY4065967 — Administered orally
  Arms: LY4065967 Part A; LY4065967 Part B; LY4065967 and Rosuvastatin Part D
Drug: Placebo — Administered orally
  Arms: Placebo Part A; Placebo Part B
Drug: Rosuvastatin — Administered orally
  Arms: LY4065967 and Rosuvastatin Part D

SUMMARY:
The purpose of this study is to obtain safety and tolerability data of the study drug known as LY4065967 and rosuvastatin in healthy Japanese participants. Blood tests will be performed to check how much LY4065967 and rosuvastatin get into the bloodstream and how long it takes the body to eliminate it. This is a 3-part study and will last approximately 2 weeks excluding screening period for each part.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants who are overtly healthy as determined by medical evaluation including medical history and physical examination
* Have a body mass index within the range 18 to 30 kilogram per square meter (kg/m2)
* Have a body weight of:
* ≥ 40 kilograms (kg) for individuals assigned female at birth
* ≥ 50 kg for individuals assigned male at birth

Exclusion Criteria:

* Have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or convulsions that, in the judgment of the investigator, indicate a medical problem that would preclude study participation
* Have an abnormality in the 12-lead echocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of clinically significant multiple or severe drug allergies or severe posttreatment hypersensitivity reactions, which in the opinion of the investigator may hamper participation in the study
* Show evidence of hepatitis C and/or have a positive hepatitis C virus antibody test
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antigen and/or antibodies.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of syphilis or have a positive syphilis test.
* Have an abnormal blood pressure (supine) as determined by the investigator
* Are pregnant or intend to become pregnant or to breastfeed during the study.
* Participants with a history of drug abuse which, in the opinion of the investigator, is clinically significant or who test positive for drugs of abuse at screening or admission
* Have alcohol intake that exceeds recommended average weekly alcohol consumption limits per local regulation, or an amount deemed significant by the investigator
* Smoke more than 10 cigarettes per day or the equivalent including electronic cigarettes
* Are unwilling to comply with the dietary restrictions required for this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered to be Related to Study Drug Administration | Baseline to 7 Days
  Part A: A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module
Part B: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered to be Related to Study Drug Administration | Baseline to 12 Days
  Part B: A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module
Part D: PK: Maximum Concentration (Cmax) of Rosuvastatin | Predose on Day 1 Through 72 Hours Post-Dose
  Part D: PK: Cmax of Rosuvastatin
Part D: PK: Area Under the Concentration Versus Time Curve (AUC) of Rosuvastatin | Predose on Day 1 Through 72 Hours Post-Dose
  Part D: PK: AUC of Rosuvastatin

SECONDARY OUTCOMES:
Part A : Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4065967 | Predose on Day 1 Through 48 Hours Post-Dose
  Part A: PK: Cmax of LY4065967
Part B: PK: Cmax of LY4065967 | Predose on Day 1 Through Day 9
  Part B: PK: Cmax of LY4065967
Part A and B: PK: Area Under the Concentration Versus Time Curve (AUC) of LY4065967 | Predose on Day 1 Through 48 Hours Post-Dose
  Part A and B: PK: AUC of LY4065967
Part D: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4065967 | Day 5 Through Day 11
  Part D: PK: Cmax of LY4065967
Part D: PK: Area Under the Concentration Versus Time Curve (AUC) of LY4065967 | Day 5 Through Day 11
  Part D: PK: AUC of LY4065967

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No